CLINICAL TRIAL: NCT03352466
Title: First-in-human, Randomized, Placebo-controlled, Double-blind, Dose-escalation Study of the Safety and Immunogenicity of NasoShield
Brief Title: NasoShield Study of Safety and Immunogenicity
Acronym: NasoShield
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: ALT201-101
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: Anthrax
MeSH Terms: conditions — Anthrax | interventions — Biothrax

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- NasoShield very low dose - 1 X 10^8 vp (Experimental): Single intranasal spray (Part A)
  Interventions: Biological: NasoShield
- NasoShield low dose - 1 X 10^9 vp (Experimental): Single intranasal spray (Part A)
  Interventions: Biological: NasoShield
- NasoShield medium dose - 1 X 10^10 vp (Experimental): Single intranasal spray (Part A)
  Interventions: Biological: NasoShield
- NasoShield high dose - Part A -1 X 10^11 vp (Experimental): Single intranasal spray (Part A)
  Interventions: Biological: NasoShield
- NasoShield high dose - Part B - 1 X 10^11 vp (Experimental): 2 intranasal sprays 21 days apart (Part B)
  Interventions: Biological: NasoShield
- Placebo (Placebo Comparator): Normal saline, single intranasal spray (Part A) or two intranasal sprays 21 days apart (Part B)
  Interventions: Other: Placebo
- BioThrax (Active Comparator): Three intramuscular injections 15 days apart (Part A)
  Interventions: Biological: BioThrax

INTERVENTIONS:
Biological: NasoShield — NasoShield is an adenovirus-vectored anthrax vaccine.
  Arms: NasoShield high dose - Part A -1 X 10^11 vp; NasoShield high dose - Part B - 1 X 10^11 vp; NasoShield low dose - 1 X 10^9 vp; NasoShield medium dose - 1 X 10^10 vp; NasoShield very low dose - 1 X 10^8 vp
Biological: BioThrax — Commercially available anthrax vaccine
  Arms: BioThrax
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
This study is a Phase 1, randomized, double-blind, placebo-controlled, dose-escalation clinical trial to evaluate the safety and immunogenicity of NasoShield in healthy adults 18 to 49 years of age.

DETAILED DESCRIPTION:
This study is a Phase 1, randomized, double-blind, placebo-controlled, dose-escalation clinical trial to evaluate the safety and immunogenicity of NasoShield in healthy adults 18 to 49 years of age. Subjects will be screened within 28 days of randomization (Day 1). The study is comprised of 2 parts:

* Part A: Approximately 120 subjects who meet all inclusion and no exclusion criteria and provide written informed consent will be enrolled into 4 sequential cohorts of 30 subjects each defined by the NasoShield dose (1×108, 1×109, 1×1010, and 1×1011 vp). Within each cohort (and the sentinel group in the first dose cohort), subjects will be randomized in a 4:1:1 ratio to receive 1 intranasal dose of NasoShield (Day 1), 1 intranasal dose of placebo (Day 1), or 3 subcutaneous 0.5 mL doses of BioThrax 14 days apart (Days 1, 15, and 29). NasoShield and placebo will be administered in a double-blind fashion, and BioThrax will be administered in an open-label fashion.
* Part B: Approximately 25 subjects who meet all inclusion and no exclusion criteria and provide written informed consent will be randomized in a 4:1 ratio to receive 2 intranasal doses of NasoShield at the highest well tolerated dose from Part A or placebo 21 days apart (Days 1 and 22). NasoShield and placebo will be administered in a double-blind fashion.

Subjects will return to the investigational site for multiple visits through Day 361. At each visit, the subject will be asked about the interim medical history and use of any medications, and safety and immunogenicity assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 to 49 years of age, inclusive
2. Good general health status as determined by the Investigator
3. Adequate venous access for repeated phlebotomies
4. Screening laboratory results within institutional normal range or Grade 1 abnormality if the Investigator documents clinical insignificance. Creatine kinase or bilirubin may be Grade 2 if associated with normal alanine aminotransferase (ALT) and aspartate aminotransferase (AST) and the Investigator considers the result not to be clinically significant due to vigorous exercise or Gilbert's syndrome
5. Negative drug and alcohol screen at Screening and predose on Day 1
6. For women who have not been surgically sterilized and do not have laboratory confirmation of postmenopausal status, negative pregnancy test
7. Willingness to practice a highly effective method of contraception: abstinence, sex only with persons of the same sex, monogamous relationship with a postmenopausal partner, monogamous relationship with vasectomized partner, vasectomy, surgical sterilization (hysterectomy, bilateral tubal ligation, salpingectomy, or oophorectomy), licensed hormonal methods, intrauterine device (IUD), or consistent use of a barrier method (eg, condom, diaphragm) with spermicide for 28 days after the last IP dose
8. Willingness to participate and comply with all aspects of the study through the entire study period, including nasopharyngeal swabs and blood and urine samples
9. Provision of written informed consent

Exclusion Criteria

1. Pregnant, possibly pregnant, or lactating women
2. Household contacts of pregnant women, children < 5 years of age, or immunocompromised individuals for the period up through 2 weeks postvaccination
3. Persons who care for pregnant women, children < 5 years of age, or immunocompromised individuals for the period up through 2 weeks postvaccination
4. Body mass index > 35.0 kg/m2
5. Positive result for HIV, hepatitis B virus, or hepatitis C virus at Screening
6. Asthma or other chronic lung disease that is greater than mild in severity. Specifically excluded are participants with any of the following events in the past year:

   * Daily symptoms
   * Daily use of short acting beta 2 agonists
   * Use of inhaled steroids or theophylline
   * Use of pulse systemic steroids
   * Emergency care or hospitalization related to asthma or other chronic lung disease
   * Systemic steroids for asthma exacerbation
7. History of diabetes mellitus (gestational diabetes is allowed if treatment was not required postpartum and serum glucose is currently in the normal range)
8. History of coronary artery disease, arrhythmia, or congestive heart failure
9. Clinically significant ECG abnormality as determined by the Investigator
10. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 95 mmHg) at Screening or predose on Day 1
11. History of anaphylaxis or angioedema
12. Known allergy to any of the ingredients in the vaccine formulation
13. Known allergy or sensitivity to latex
14. History of chronic rhinitis, nasal septal defect, cleft palate, nasal polyps, or other nasal abnormality that might affect vaccine administration
15. Previous nasal surgery or nasal cauterization
16. Any symptoms of upper respiratory infection or temperature > 38°C within 3 days before Day 1
17. Any symptoms within 24 hours before Day 1 of upper respiratory illness or allergy flare-up that, in the opinion of the Investigator, presents as nasal congestion or rhinorrhea that could inhibit the proper administration of the IP
18. Known or suspected malignancy, excluding non-melanoma skin cancers and other early stage surgically excised malignancies that the Investigator considers to be exceedingly unlikely to recur
19. Immunocompromised individuals, including those who have used corticosteroids (including intranasal steroids), alkylating drugs, antimetabolites, radiation, immune-modulating biologics, or other immunomodulating therapies within 90 days before Day 1 or those who plan use during the study period
20. Use of statin medication within 30 days before Day 1 (see list in Section 6.8.1)
21. Receipt of intranasal medications (including over-the-counter medications) within 30 days before Day 1
22. Receipt of any IP within 30 days before Day 1
23. Receipt of any vaccine within 30 days before Day 1
24. Receipt of intranasal vaccine within 90 days before Day 1
25. Receipt of any licensed or investigational anthrax vaccine
26. Any change in medication for a chronic medical condition within 30 days before Day 1
27. Past regular use or current use of intranasal illicit drugs
28. Smokers, including smoking of any type (eg, cigarettes, electronic cigarettes, marijuana). Prior smokers must have quit smoking at least 30 days before Day 1.
29. Any medical, psychiatric, or social condition or occupational or other responsibility that in the judgment of the Investigator would interfere with or serve as a contraindication to protocol adherence, assessment of safety (including reactogenicity), or a subject's ability to give informed consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Reactogenicity | For 14 days after vaccination
  Subjects will record solicited local and systemic events for 14 days after each dose
Adverse events (AEs) | From Day 1 to Day 361
  All adverse events from Day 1 to Day 57, SAEs, medically attended AEs and new onset chronic illnesses Day 1 to Day 361

SECONDARY OUTCOMES:
Anti-PA immunoglobulin G (IgG) | From Day 1 to Day 361
  Titer measured by enzyme-linked immunosorbent assay (ELISA) in serum
Toxin neutralization assay (TNA) | From Day 1 to Day 361
  50% neutralization factor (NF50) titer measured by cytotoxic assay in serum

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel DeNoia, MD, Principal Investigator — ICON plc
Locations (2):
- United States (2):
  - Optimal Research, LLC, Melbourne, Florida
  - ICON Early Phase Services, LLC, San Antonio, Texas